CLINICAL TRIAL: NCT00603395
Title: A Prospective Clinical Study On A Total Hip Resurfacing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anna Ziekenhuis, Geldrop, Netherlands (Other)
Responsible Party: Principal Investigator, Walter van der Weegen, Researcher, St. Anna Ziekenhuis, Geldrop, Netherlands
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-6
Record Dates: First submitted 2007-12-23; First posted 2008-01-29 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Arthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReCap (Other): ReCap Total Hip Resurfacing System
  Interventions: Device: ReCap Total Hip Resurfacing System

INTERVENTIONS:
Device: ReCap Total Hip Resurfacing System — This is a hip resurfacing system.

SUMMARY:
This prospective clinical study is to demonstrate the efficacy and safety of ReCap Total Hip Resurfacing System.

ELIGIBILITY:
Inclusion Criteria:

* intended for skeletally mature individuals undergoing primary surgery as a result of hip degenerative joint disease, or any composite diagnoses, including:

  * Osteoarthritis
  * Avascular necrosis
  * Traumatic arthritis
  * Legg Perthes
  * Rheumatoid arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2004-09; Primary Completion 2012-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score, Device Revision/Removal, Radiographic Evaluation | 2 years postoperative

SECONDARY OUTCOMES:
Complications | Anytime

CONTACTS AND LOCATIONS:
Overall Officials: H J Hoekstra, MD, Principal Investigator — St. Anna hospital, Geldrop; T Sybesma, PhD, Principal Investigator — St. Anna hospital, Geldrop
Locations (1):
- Knowledge Center for Orthopedic Surgery, St. Anna hospital, Geldrop, Netherlands

REFERENCES:
- [Derived] van der Weegen W, Hoekstra HJ, Sijbesma T, Austen S, Poolman RW. Hip resurfacing in a district general hospital: 6-year clinical results using the ReCap hip resurfacing system. BMC Musculoskelet Disord. 2012 Dec 13;13:247. doi: 10.1186/1471-2474-13-247. PMID 23234268